CLINICAL TRIAL: NCT07198529
Title: Optical Coherence Tomography for Stent Optimization and Its Impact on Short-Duration Dual Antiplatelet Therapy: A Single-Center, Prospective, Exploratory Study
Brief Title: OCT-Guided Stent Optimization for Short-Duration Dual Antiplatelet Therapy in Stable Angina
Acronym: COMFORT-SHORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Park, Soohyung, Assistant Professor, Interventional Cardiologist, Korea University Guro Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No.2025GR0393; KOR-2023-02 (Other Grant/Funding Number: Abott)
Record Dates: First submitted 2025-09-19; First posted 2025-09-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stable Angina; Coronary Artery Disease
Keywords: Optical coherence tomography; stable angina; dual antiplatelet therapy; stent optimization; percutaneous coronary intervention
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, open-label study with a parallel assignment design. All patients undergo OCT-guided PCI. Based on OCT findings, patients are categorized into two groups: those with optimized stent results receive short-duration DAPT (1 month), while those with suboptimal stent results continue standard DAPT (6-12 months) according to guidelines. Outcomes will be compared between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Short DAPT (Experimental): Patients with optimized stent results confirmed by OCT will receive 1 month of dual antiplatelet therapy followed by clopidogrel monotherapy.
  Interventions: Drug: Short DAPT; Device: OCT-guided PCI
- Standard DAPT (Active Comparator): Patients with suboptimal stent results (malapposition, dissection, under-expansion) with high bleeding risk will continue dual antiplatelet therapy for 6 months, according to guideline recommendations.
  Interventions: Drug: Standard DAPT; Device: OCT-guided PCI
- Extended DAPT (Active Comparator): Patients with suboptimal stent results and high ischemic risk, as judged by the operator, will remain on dual antiplatelet therapy for 12 months.
  Interventions: Drug: Extended DAPT; Device: OCT-guided PCI

INTERVENTIONS:
Drug: Short DAPT — Patients receive aspirin and clopidogrel for 1 month after PCI. After 1 month, aspirin is discontinued and clopidogrel monotherapy is continued.
  Arms: Short DAPT
Drug: Standard DAPT — Patients with high bleeding risk will receive aspirin and clopidogrel for 6 months after PCI (unoptimization confirmed in OCT), followed by single antiplatelet therapy thereafter.
  Arms: Standard DAPT
Drug: Extended DAPT — Patients (with stet unoptimazation results in OCT imaging) receive aspirin and clopidogrel for 12 months after PCI.
  Arms: Extended DAPT
Device: OCT-guided PCI — All patients undergo percutaneous coronary intervention with mandatory intravascular imaging using optical coherence tomography to assess stent optimization (expansion, apposition, dissection).

SUMMARY:
This study aims to evaluate whether the use of optical coherence tomography (OCT), an advanced intravascular imaging tool, can improve stent implantation results and make it possible to shorten the duration of dual antiplatelet therapy (DAPT) in patients with stable angina who undergo percutaneous coronary intervention (PCI).

PCI with drug-eluting stents is a standard treatment for patients with stable angina, and these patients are usually prescribed DAPT for 6 to 12 months to prevent stent thrombosis and other complications. However, extended use of DAPT increases the risk of bleeding, which can lead to significant medical problems, especially in patients with high bleeding risk.

OCT provides detailed, high-resolution images of the coronary arteries and the implanted stents, allowing physicians to optimize stent expansion and positioning. By ensuring that the stent is well-placed and fully expanded, OCT guidance may lower the risk of complications, potentially reducing the need for prolonged DAPT.

In this prospective study, patients with stable angina who require stent implantation will be enrolled and treated with OCT-guided PCI followed by a short course of DAPT. Their outcomes will be compared with those managed using conventional strategies.

The primary goal of this trial is to determine whether OCT-guided stent optimization can safely support a short-duration DAPT strategy, thereby reducing bleeding risk without compromising protection against ischemic events such as restenosis, myocardial infarction, or stent thrombosis.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) remains one of the leading causes of death worldwide, and more than 80% of deaths from coronary artery disease (CAD) occur in individuals aged 65 years or older. Elderly patients often have multiple comorbidities, such as diabetes mellitus, hypertension, and chronic kidney disease, which increase both ischemic and bleeding risks. For these patients, the management of dual antiplatelet therapy (DAPT) after percutaneous coronary intervention (PCI) is particularly challenging, as physicians must balance ischemic protection against the risk of bleeding complications.

Optical coherence tomography (OCT) provides high-resolution intravascular imaging that allows precise assessment of stent apposition, expansion, and the presence of dissections. Previous studies, including Kubo et al. (2022), have proposed OCT-based criteria for stent optimization, demonstrating that inadequate stent expansion or a minimum lumen area (MLA) < 4.5 mm² is associated with worse outcomes. However, to date, few clinical studies have directly evaluated whether OCT-guided stent optimization can support individualized adjustment of DAPT duration.

The COMFORT-SHORT study is a prospective, single-center, open-label pilot registry designed to investigate the safety and feasibility of OCT-guided stent optimization in applying short-term DAPT strategies. Patients with stable angina undergoing PCI with drug-eluting stent implantation will be enrolled. All participants will undergo OCT during PCI to evaluate stent deployment. Stent size and length will be determined based on OCT analysis, and final imaging will be reviewed to confirm whether the procedure meets predefined optimization criteria.

Patients whose stents are confirmed as optimized will be transitioned to 1 month of DAPT followed by clopidogrel monotherapy. Patients with suboptimal results (e.g., malapposition, medial dissection, under-expansion) will continue standard DAPT for 6-12 months, based on guideline recommendations and individual bleeding. Importantly, patients with non-optimized stents will not be excluded; they will be followed prospectively, and outcomes will be compared with those of optimized patients.

The primary endpoint is the incidence of net adverse clinical events (NACE) at 12 months, comparing short-term versus standard DAPT strategies according to stent optimization status. All enrolled patients will undergo scheduled follow-up at 1, 6, and 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo PCI using a cobalt-chromium everolimus-eluting stent (CoCr-EES)
* Diagnosis of stable angina
* Ability and willingness to provide written informed consent approved by the Institutional Review Board (IRB), and to comply with the study protocol and clinical follow-up schedule
* Age ≥ 19 years

Exclusion Criteria:

* Patients diagnosed with acute coronary syndrome (ACS), including unstable angina or acute myocardial infarction
* Contraindications to antiplatelet therapy or OCT imaging
* Presence of lesions with severe stenosis, heavy calcification, or marked vessel tortuosity that prevent passage of a guidewire or catheter
* Patients with previously implanted coronary stents in the target lesion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Cardiovascular Events (NACE) | 12 months after the index PCI
  Composite of cardiac death, non-fatal myocardial infarction, definite/probable stent thrombosis (ARC definition), stroke, repeat coronary revascularization, or clinically significant bleeding defined as BARC types 2, 3, or 5. Analyses will use time-to-first-event; each component will also be summarized separately as secondary outcomes per protocol.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 12 months after PCI
  Composite of cardiac death, non-fatal myocardial infarction, definite/probable stent thrombosis (ARC), repeat coronary revascularization, or stroke (time-to-first-event).
All bleeding events | 12 months after the index PCI
  Any bleeding by BARC criteria (types 1-5).
All-cause death | 12 months after the index PCI
  Death from any cause.
Cardiac death | 12 months after the index PCI
  Death due to cardiac causes (e.g., MI, sudden cardiac death, heart failure), per protocol definition.
Myocardial infarction | 12 months after the index PCI
  MI defined per protocol-specified criteria (e.g., Fourth Universal Definition of MI); adjudicated events will be counted.
Stent thrombosis | 12 months
  Definite or probable stent thrombosis per ARC definitions.
Repeat revascularization | 12 months
  Any coronary revascularization (PCI or CABG), including TLR/TVR as defined in the protocol.
Stroke | 12 months
  Ischemic or hemorrhagic stroke confirmed by clinical assessment and/or neuroimaging, with a new focal neurologic deficit lasting >24 hours or resulting in death.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Center, Department of Internal Medicine, Korea University Guro Hospital, Seoul, Gurodong-ro, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing may be considered after study completion and publication of the main results, depending on institutional policies and participant privacy considerations.